CLINICAL TRIAL: NCT05105724
Title: Clinical Study of Ovarian Injection of Autologous Platelet-rich Plasma to Improve Responsiveness and Embryo Quality in Patients With Poor Ovarian Response
Brief Title: Autologous Platelet-rich Plasma to Improve Responsiveness and Embryo Quality in Patients With Poor Ovarian Response
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing University (Other)
Responsible Party: Principal Investigator, Li-jun Ding, Principal Investigator of Reproductive Medicine Center of The Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SZ-2019-PRP
Record Dates: First submitted 2021-10-10; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP (Experimental): ovarian injections of PRP were administered to the patients
  Interventions: Biological: PRP
- No ovarian puncture or injection (No Intervention): no ovarian puncture or injection was used in the patients

INTERVENTIONS:
Biological: PRP — PRP was prepared using double centrifugation of the patient's autologous whole blood, and 400 µL of PRP was injected via vaginal puncture into the ovarian parenchyma.
  Arms: PRP

SUMMARY:
This study was a prospective randomized controlled trial. Patients with POR who were aged <40 years and underwent IVF/ICSI with assisted ovulation induction at our hospital were enrolled in the study. After randomization using Excel (Microsoft Corporation, Albuquerque, NM, USA), these patients were divided into two groups. Group A was the experimental group, wherein ovarian injections of PRP were administered to the patients, and group B was the control group, wherein no ovarian puncture or injection was used in the patients.

DETAILED DESCRIPTION:
Poor ovarian response (POR) is a pathological state, wherein the ovaries are insensitive to exogenous gonadotropin (Gn) stimulation; it is often noted older populations with ovarian hypofunction. POR mainly manifests as the development of only few follicles during ovarian stimulation cycles, low peak levels of blood estrogen on human chorionic Gn (HCG) trigger day, high dosage of exogenous Gn, high rates of cycle cancellation, low number of oocytes retrieved, and low rates of clinical pregnancy. The incidence of POR during ovulation induction in assisted reproduction is reported to be approximately 9%-24%. With the increasing age of individuals at marriage and childbearing as well as the reform of the national family planning policy, an increasing number of women of advanced maternal age have resorted to assisted reproductive technology for fertility, resulting in an increased proportion of patients with POR in China. Repeated in-vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) cycles and adverse pregnancy outcomes of patients with POR have undoubtedly resulted in great financial burden and psychological pressure on infertile couples. Therefore, the individualized selection of an appropriate ovulation induction protocol has become a key factor in terms of improving ovarian responsiveness, which can in turn improve ovarian sensitivity to ovulation drugs and increase oocyte quantity and quality when the patient is supplemented with pre-treatment prior to ovulation induction.

The intraperitoneal injection of autologous platelet-rich plasma (PRP) into the ovaries of mice of the cyclophosphamide-induced premature ovarian failure model resulted in an increase in ovarian cortical volume, preantral follicle number, and antral follicle and their corresponding oocyte diameters. This finding suggests that PRP has a positive effect on the tissue repair of damaged ovaries and that it stimulates the growth of various follicles after ovarian damage in animals, is involved in oogenesis, induces an increase in the number of follicles and granulosa cells, and stimulates estrogen secretion. The addition of PRP to in-vitro three-dimensional cultures of follicles increases the viability and growth of human primordial and preantral follicles and produced more beneficial growth factors. The Pantos team pioneered the administration of intra-ovarian injections of PRP to four infertile patients of advanced maternal age with ovarian hypofunction. These patients' ovarian reserves improved, as evidenced by their elevated serum anti-Müllerian hormone (AMH) levels, decreased follicle-stimulating hormone (FSH) levels, and/or increased total antral follicular counts. Then, the patients received IVF treatment, each patient receiving at least one blastocyst for cryopreservation. A recent clinical study used PRP in 19 patients with POR. Two of these patients had spontaneous pregnancies and one had a successful clinical pregnancy. Taken together, this evidence suggests the promising use of PRP in ovarian tissue and the potential of PRP as a novel effective treatment option for patients with POR.

In light of the current situation of POR treatment, the investigators proposed a clinical research project of ovarian injection of autologous PRP for the treatment of POR. The PRP used clinically has been evaluated in well-developed preclinical safety studies and necessary quality control without any ethical controversy. Moreover, PRP does not pose a medical risk and has high safety levels in the treatment of diseases. The goal of our project was to aid in the development of new methods of POR treatment that can meet the urgent fertility needs of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥20 years and <40 years;
2. Underwent at least one IVF/ICSI ovulation induction cycle at our center and with a number of retrieved oocytes of ≤3;
3. Total antral follicular count of <5-7 or AMH levels of <0.5-1.1 μg/L.

Exclusion Criteria:

1. Chromosomal abnormalities in either parent;
2. Acute infectious diseases, endocrine metabolic diseases, and other such conditions;
3. Underwent surgery for borderline ovarian cancer or malignant tumors;
4. Abnormal uterine development, uterine adhesions, or other untreated endometrial lesions;
5. Factors affecting oocyte retrieval or ovarian injections, such as ovarian cysts of ≥3 cm, ovarian endometriosis cysts, severe pelvic adhesions, and poor visualization of ovarian positions;
6. Conditions affecting the pregnancy outcome, such as untreated hydrosalpinx, hysteromyoma of ≥4 cm, adenomyosis, and stage III-IV endometriosis;
7. Azoospermia or severe oligospermia and teratozoospermia in the male partner;
8. Participated in another investigational trial within the previous year;
9. Allergies to blood products.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-20 (Actual); Primary Completion 2022-07-20 (Estimated); Study Completion 2022-07-20 (Estimated)

PRIMARY OUTCOMES:
number of oocytes retrieved | 30 days after PRP injected
  When at least one dominant follicle reached a diameter of 18 mm or higher, 0.2 mg triptorelin was combined with 1,000 U HCG as the trigger, and ovarian puncture was performed 36 hours later for oocyte retrieval. The number of oocytes retrieved was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Haixiang Sun, PhD, Study Director — The affiliated Drum Towel Hospital of Nanjing University Medical School
Locations (1):
- Reproductive Medicine Center, The affiliated Drum Towel Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China